CLINICAL TRIAL: NCT04116242
Title: MERTK Signalling in Monocytes/Macrophages in Patients With Liver Disease
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: EKSG 15/074; me19Bernsmeier2
Record Dates: First submitted 2019-10-03; First posted 2019-10-04 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Liver Disease; Cirrhosis of the Liver; Acute-On-Chronic Liver Failure; Liver Failure
Keywords: immunoparesis; monocyte dysfunction; MER receptor tyrosine kinase (MERTK); innate immune dysfunction; circulating monocytes/macrophages; MERTK signalling
MeSH Terms: conditions — Liver Diseases; Fibrosis; Acute-On-Chronic Liver Failure; Liver Failure | interventions — Blood Specimen Collection; Hepatectomy; Urination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biological material will be stored in -80°C and -140°C freezers at the sites of recruitment.
  If biological material (e.g. liver biopsies, liver resections, ascites, urine, gut biopsies) are sampled routinely for clinical reasons and exceeding material allows additional scientific investigations, a small amount of the material will be used. The samples will be destroyed 10 years after publication of the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- cirrhosis of the liver, stadium Child A: sampling of biological material and health related data collection longitudinally in 6-monthly intervals up to 36 months
  Interventions: Other: blood sampling for research purpose; Other: clinical data collection; Other: Health-related Questionnaires; Other: Sampling other biological materials (e.g. liver biopsies, liver resections, ascites, urine, gut biopsies)
- cirrhosis of the liver, stadium Child B: sampling of biological material and health related data collection longitudinally in 6-monthly intervals up to 36 months
  Interventions: Other: blood sampling for research purpose; Other: clinical data collection; Other: Health-related Questionnaires; Other: Sampling other biological materials (e.g. liver biopsies, liver resections, ascites, urine, gut biopsies)
- cirrhosis of the liver, stadium Child C: sampling of biological material and health related data collection longitudinally in 6-monthly intervals up to 36 months
  Interventions: Other: blood sampling for research purpose; Other: clinical data collection; Other: Health-related Questionnaires; Other: Sampling other biological materials (e.g. liver biopsies, liver resections, ascites, urine, gut biopsies)
- cirrhosis of the liver, acutely decompensated: sampling of biological material and health related data collection on days 1 (Baseline), 3, 7, and 14. If acutely decompensated patients re-compensate they will be followed 6-monthly for up to 36 months
  Interventions: Other: blood sampling for research purpose; Other: clinical data collection; Other: Health-related Questionnaires; Other: Sampling other biological materials (e.g. liver biopsies, liver resections, ascites, urine, gut biopsies)
- acute liver failure: sampling of biological material and health related data collection on days 1 (Baseline), 3, 7, and 14. If acutely decompensated patients re-compensate they will be followed 6-monthly for up to 36 months
  Interventions: Other: blood sampling for research purpose; Other: clinical data collection; Other: Health-related Questionnaires; Other: Sampling other biological materials (e.g. liver biopsies, liver resections, ascites, urine, gut biopsies)
- healthy controls: sampling of biological material and health related data collection on day 1 (Baseline)
  Interventions: Other: blood sampling for research purpose; Other: clinical data collection; Other: Health-related Questionnaires

INTERVENTIONS:
Other: blood sampling for research purpose — blood sampling for research purpose (about 30ml) taken by venepuncture or from intravenous catheters if already in place
Other: clinical data collection — clinical data collection in order to document the stage of disease, the presence of infection and existing complications of cirrhosis (ascites, hepatic encephalopathy, renal dysfunction, pulmonary dysfunction) and concomitant disease. These data will be collected for clinical reasons as highly important in the context of patients with cirrhosis and possible decompensation or liver failure and will therefore not require additional time
Other: Health-related Questionnaires — Health-related Questionnaires (Questionnaire_CLD) regarding sleep characteristics (Pittsburgh sleep Quality index, PSQI), daytime sleepiness (Epworth sleepiness scale, ESS), anxiety and depression (Hospital Anxiety and Depression Scale, HADS) and quality of life (EQ-5D-5L)
Other: Sampling other biological materials (e.g. liver biopsies, liver resections, ascites, urine, gut biopsies) — Other biological material (e.g. liver biopsies, liver resections, ascites, urine, gut biopsies) will only be investigated if sampled for clinical reasons and if excessive material is available that is not needed for clinical purpose.
  Groups: acute liver failure; cirrhosis of the liver, acutely decompensated; cirrhosis of the liver, stadium Child A; cirrhosis of the liver, stadium Child B; cirrhosis of the liver, stadium Child C

SUMMARY:
This study is to investigate MER receptor tyrosine kinase (MERTK) signalling cascade on monocytes and tissue macrophages in respect to innate immune function of the cells in patients with cirrhosis at different stages of disease (Child A, B, C, acute decompensation, acute-on-chronic liver failure (ACLF)) and in comparison to patients with acute liver failure and to healthy controls.

DETAILED DESCRIPTION:
MER receptor tyrosine kinase (MERTK) signalling cascade becomes activated on monocytes/macrophages during disease progression of liver cirrhosis from Child Pugh A to B/C, corresponding to early stages of decompensation, and before the receptor expression is increased. Factors involved in activation of the MERTK signalling cascade might be microbial products such as bacterial deoxyribonucleic acid (DNA) and other toll-like receptor (TLR)-ligands, MERTK ligands and cytokines, as shown elevated in cirrhotic patients.

Given the observation that MERTK levels peak on the day of admission with organ failure and decrease in patients surviving the episode of acute-on-chronic liver failure (ACLF), MERTK Inhibition at a time during progression of cirrhosis but before manifestation of acute decompensation with no cirrhosis (AD) or ACLF might prevent infectious complications, decompensation and improve survival in patients with cirrhosis.

This study is to investigate MER receptor tyrosine kinase (MERTK) signalling cascade on monocytes and tissue macrophages in respect to innate immune function of the cells in patients with cirrhosis at different stages of disease (Child A, B, C, acute decompensation, acute-on-chronic liver failure (ACLF)) and in comparison to patients with acute liver failure and to healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Patients with compensated or decompensated chronic liver disease
* Patients with acute- or acute-on-chronic chronic liver failure
* Controls with no liver disease

Exclusion Criteria:

* Evidence of disseminated malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Prospective recruitment of patients with cirrhosis, acute decompensation, acute liver failure as pathological controls and healthy controls or controls with no liver disease at the Cantonal Hospital St. Gallen (KSSG), University Hospital Basel, St. Mary's Hospital, Imperial College London and King's College Hospital, London, UK.
Sampling Method: Probability Sample
Enrollment: 277 (Actual)
Dates: Start 2015-08-27 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-06-10 (Actual)

PRIMARY OUTCOMES:
Change in MERTK signalling cascade on monocytes | days 1 (Baseline), 3, 7, and 14; then followed 6-monthly for up to 36 months
  Change in MERTK signalling cascade on monocytes in respect to innate immune function of the cells in patients with cirrhosis at different stages of disease (Child A, B, C, acute decompensation, ACLF) and in comparison to patients with acute liver failure and to healthy controls
Change in MERTK signalling cascade on tissue macrophages | days 1 (Baseline), 3, 7, and 14; then followed 6-monthly for up to 36 months
  Change in MERTK signalling cascade on tissue macrophages in respect to innate immune function of the cells in patients with cirrhosis at different stages of disease (Child A, B, C, acute decompensation, ACLF) and in comparison to patients with acute liver failure and to healthy controls

SECONDARY OUTCOMES:
Change in mechanism of MERTK activation in cell culture models using monocytes | days 1 (Baseline), 3, 7, and 14; then followed 6-monthly for up to 36 months
  Change in mechanism of MERTK activation in cell culture models using healthy and diseased monocytes in vitro and ex vivo

CONTACTS AND LOCATIONS:
Overall Officials: Christine Bernsmeier, PD Dr. Dr., Principal Investigator — Universitätsspital Basel, Departement Biomedizin, Gastroenterologie und Hepatologie
Locations (4):
- Switzerland (2):
  - University Hospital Basel, Hepatology Department and Laboratory, Basel
  - Cantonal Hospital St. Gallen, Sankt Gallen
- United Kingdom (2):
  - King's College Hospital, Institute of Liver studies, London
  - St. Mary's Hospital, Imperial College London, Section of Hepatology, London